CLINICAL TRIAL: NCT05077943
Title: The Effect of Home-based Breathing and Chest Mobilisation Exercise on Cardiorespiratory Functional Capacity of Covid-19 Survivor With Cardiovascular Comorbidity
Brief Title: The Effect of Home-based Exercise on Functional Capacity of Covid-19 Survivor With Cardiovascular Comorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Bambang Dwiputra, MD, MD Cardiologist, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Home based Exercise PostCovid
Record Dates: First submitted 2021-09-29; First posted 2021-10-14 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Breathing Exercise; Cardiovascular Diseases
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases | interventions — Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Breathing Exercise (Active Comparator): Patients will do the second phase of cardiac rehabilitation for minimum 5 times per week, 30 minutes each time, in 3 months without being supervised
  Interventions: Behavioral: Second phase cardiac rehabilitation
- With Breathing Exercise (Experimental): Patients will do the second phase of cardiac rehabilitation for minimum 5 times per week, 30 minutes each time and breathing and chest mobilization exercise for 3 times per week. They will be supervised through online meetings.
  Interventions: Behavioral: Breathing and chest mobilization exercises

INTERVENTIONS:
Behavioral: Breathing and chest mobilization exercises — Patients walk regularly 5 times per week and increase the distance day by day according to their improved ability. Patients also do breathing and chest mobilization exercise 3 times per week. It is a recorded moderated exercise for 30 minutes duration. Patients can access the video as a home-based activity through an online videos platform and will be supervised.
  Arms: With Breathing Exercise
Behavioral: Second phase cardiac rehabilitation — Independently, patients walk regularly 5 times per week and increase the distance day by day according to their improved ability without breathing and chest mobilization exercise.
  Arms: No Breathing Exercise

SUMMARY:
Objective propose: to investigate the effect of home based breathing exercise and chest mobilization on the cardiorespiratory functional capacity of Covid-19 survivors with cardiovascular comorbidity.

Breathing exercise and chest mobilization are proven to increase lung functional capacity in Covid-19 survivors. It is hypothesized that breathing exercise and chest mobilization in Covid-19 survivors will give benefits to Covid-19 survivors with cardiovascular disease.

DETAILED DESCRIPTION:
Lung restrictive disorder is one of the reasons that induce chronic fatigue in COVID-19 (Corona Virus Disease-19) survivors. It also gives a significant effect on cardiovascular patients who are in the second phase of cardiac rehabilitation. Breathing exercise and chest mobilization are proven to increase lung functional capacity in Covid-19 survivors. On the other hand, there is still no research that shows the effectiveness of Breathing exercises and chest mobilization in Covid-19 survivors who are suffering from cardiovascular problems.

Patients in National Cardiac Center Hospital, Jakarta, with a history of Covid-19 and have cardiovascular disease are recruited. They will undergo pre and post-exercise examinations such as blood sampling, do 6 minutes walking test, Peak Cough Flow and Peak Flow Rate test, measuring the chest dimension, treadmill, and answer the European Quality of Life Five Dimension (EQ-5D) questions. With randomization, patients will be determined to treatment or control group. They will be prepared about what exercises should they do at home. Subjects will be supervised digitally and regularly through Zoom meetings. Exercises will be done for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who got infected by Covid-19 in 3 months before recruitment and suffering cardiovascular disease
* Able to communicate and operate Youtube and Zoom.

Exclusion Criteria:

* Limitation to move any part of the body that causes the inability to do the instructed exercise.
* Feel pain in extremities (visual analog scale >3)
* Chronic Obstructive Pulmonary Disease
* Neuromuscular disorder (stroke, peripheral neuropathy with significant motoric control disturbance
* Musculoskeletal disorder (fracture, post amputation, severe arthritis in support joints)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change of Peak Cough Flow (PC) | Change from Baseline Peak Cough Flow (PC) at 3 months
  to define the functional capacity. Unit of measure : L/min.
Change of Peak Flow Rate (PFR) | Change from Baseline Peak Flow Rate (PFR) at 3 months
  to define the functional capacity. Unit of measure : L/min.
Change of Cardiac Exercise Test | Change from Baseline Cardiac Exercise Test at 3 months
  Patients walk on treadmill. Unit of measure : minutes, METs (Metabolic Equivalent of Task)
Change of 6-minutes walking test | Change from Baseline 6-minutes walking test at 3 months
  To define initial ability to walk in 30 minutes for second phase cardiac rehabilitation (aerobic exercise). Unit of measure : meter

SECONDARY OUTCOMES:
Change of Hemoglobin | Change from Baseline Hemoglobin at 3 months
  Hemoglobin (g/dL)
Change of Hematocrit | Change from Baseline Hematocrit at 3 months
  Hematocrit (%)
Change of Erythrocyte | Change from Baseline Erythrocyte at 3 months
  Erythrocyte (million/µL)
Change of Mean Corpuscular Volume | Change from Baseline Mean Corpuscular Volume at 3 months
  Mean Corpuscular Volume (fL)
Change of Mean Corpuscular Hemoglobin | Change from Baseline Mean Corpuscular Hemoglobin at 3 months
  Mean Corpuscular Hemoglobin (pg)
Change of Mean Corpuscular Hemoglobin Concentration | Change from Baseline Mean Corpuscular Hemoglobin Concentration at 3 months
  Mean Corpuscular Hemoglobin Concentration (%)
Change of Red Cell Distribution Width | Change from Baseline Red Cell Distribution Width at 3 months
  Red Cell Distribution Width (%)
Change of Leucocyte | Change from Baseline Leucocyte at 3 months
  Leucocyte (/µL)
Change of Platelet | Change from Baseline Platelet at 3 months
  Platelet (thousand/µL)
Change of European Quality of Life Five Dimension (EQ-5D) | Change from Baseline EQ-5D at 3 months
  1=have no problem, 2=have slight problem, 3=moderate problem, 4=severe problem, 5=unable to do. We will compare the points between pre and post exercise and looking the improvement.
Change of Basophil | Change from Baseline Basophil at 3 months
  Basophil (/µL)
Change of Eosinophil | Change from Baseline Eosinophil at 3 months
  Eosinophil (/µL)
Change of Neutrophil | Change from Baseline Neutrophil at 3 months
  Neutrophil (/µL)
Change of Lymphocyte | Change from Baseline Lymphocyte at 3 months
  Lymphocyte (/µL)
Change of Monocyte | Change from Baseline Monocyte at 3 months
  Monocyte (/µL)
Change of C-Reactive Protein | Change from Baseline C-Reactive Protein at 3 months
  to determine infection markers. Unit of measure : mg/L
Change of D-dimer | Change from Baseline D-dimer at 3 months
  Unit of measure : ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Dwiputra, MD, FIHA, Principal Investigator — National Cardiovascular Center Harapan Kita Hospital Indonesia
Locations (1):
- National Cardiovascular Center Harapan Kita Hospital Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. WHO Indonesia. Coronavirus Disease 2019 (COVID-19) Situation Report-36. [Internet]. WHO; [2020 Dec 2; cited 2021 Feb 12]. Available from: https://www.who.int/indonesia/news/novel-coronavirus/situation-reports
- [Background] Halpin SJ, McIvor C, Whyatt G, Adams A, Harvey O, McLean L, Walshaw C, Kemp S, Corrado J, Singh R, Collins T, O'Connor RJ, Sivan M. Postdischarge symptoms and rehabilitation needs in survivors of COVID-19 infection: A cross-sectional evaluation. J Med Virol. 2021 Feb;93(2):1013-1022. doi: 10.1002/jmv.26368. Epub 2020 Aug 17. PMID 32729939
- [Background] Eapen MS, Lu W, Gaikwad AV, Bhattarai P, Chia C, Hardikar A, Haug G, Sohal SS. Endothelial to mesenchymal transition: a precursor to post-COVID-19 interstitial pulmonary fibrosis and vascular obliteration? Eur Respir J. 2020 Oct 15;56(4):2003167. doi: 10.1183/13993003.03167-2020. Print 2020 Oct. PMID 32859681
- [Background] Abdullahi A. Safety and Efficacy of Chest Physiotherapy in Patients With COVID-19: A Critical Review. Front Med (Lausanne). 2020 Jul 21;7:454. doi: 10.3389/fmed.2020.00454. eCollection 2020. PMID 32793618
- [Background] Sardari A, Tabarsi P, Borhany H, Mohiaddin R, Houshmand G. Myocarditis detected after COVID-19 recovery. Eur Heart J Cardiovasc Imaging. 2021 Jan 1;22(1):131-132. doi: 10.1093/ehjci/jeaa166. No abstract available. PMID 32462177
- [Background] Salman D, Vishnubala D, Le Feuvre P, Beaney T, Korgaonkar J, Majeed A, McGregor AH. Returning to physical activity after covid-19. BMJ. 2021 Jan 8;372:m4721. doi: 10.1136/bmj.m4721. No abstract available. PMID 33419740
- [Background] Ogura A, Izawa KP, Tawa H, Kureha F, Wada M, Harada N, Ikeda Y, Kimura K, Kondo N, Kanai M, Kubo I, Yoshikawa R, Matsuda Y. Impact of the COVID-19 pandemic on phase 2 cardiac rehabilitation patients in Japan. Heart Vessels. 2021 Aug;36(8):1184-1189. doi: 10.1007/s00380-021-01783-5. Epub 2021 Jan 29. PMID 33512598
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] 9. ESC. Recommendations on how to provide cardiac rehabilitation activities during the COVID-19 pandemic. [Internet] France: European Society of Cardiology; [2020 Apr 8; cited in 2021 Feb 12]. Available from: https://www.escardio.org/Education/Practice-Tools/CVD-prevention-toolbox/recommendations-on-how-to-provide-cardiac-rehabilitation-activities-during-the-c
- [Derived] Dwiputra B, Ambari AM, Triangto K, Supriami K, Kesuma TW, Zuhdi N, Phowira J, Radi B. The home-based breathing and chest mobility exercise improves cardiorespiratory functional capacity in long COVID with cardiovascular comorbidities: a randomized study. BMC Cardiovasc Disord. 2024 Oct 18;24(1):574. doi: 10.1186/s12872-024-04196-0. PMID 39425012